CLINICAL TRIAL: NCT07022821
Title: Comparison of Different Doses of Dexmedetomidine in Combination With Ketamine for Control of Post-Operative Pain in Lower Segment Caesarean Section Surgeries
Brief Title: Comparison of Dexmedetomidine + Ketamine for Postoperative Pain in C-Section
Acronym: KETODEX-CS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fatima Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Naeem, Principal Investigator, Fatima Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMH-KETODEX-CS-2025
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain; Cesarean Section Pain
Keywords: Cesarean Pain; Multimodal Analgesia; Spinal Anesthesia; Dexmedetomidine; Ketamine; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Dose Dexmedetomidine (Experimental): Dexmedetomidine 0.2 µg/kg/hr + Ketamine 0.25 mg/kg/hr infusion
  Interventions: Drug: Dexmedetomidine; Drug: ketamine
- Medium-Dose Dexmedetomidine (Experimental): Dexmedetomidine 0.3 µg/kg/hr + Ketamine 0.25 mg/kg/hr infusion
  Interventions: Drug: Dexmedetomidine; Drug: ketamine
- High-Dose Dexmedetomidine (Experimental): Dexmedetomidine 0.4 µg/kg/hr + Ketamine 0.25 mg/kg/hr infusion
  Interventions: Drug: Dexmedetomidine; Drug: ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion at one of the following doses:
  Group A: 0.2 µg/kg/hr Group B: 0.3 µg/kg/hr Group C: 0.4 µg/kg/hr Route of Administration: Intravenous Frequency: Continuous infusion during postoperative period
Drug: ketamine — Ketamine infusion at a fixed dose of 0.25 mg/kg/hr administered in all three groups.
  Route of Administration: Intravenous Frequency: Continuous infusion during postoperative period

SUMMARY:
This study aims to compare three different doses of dexmedetomidine, when combined with a fixed dose of ketamine, for pain control in women undergoing cesarean section. The goal is to find the most effective combination with the fewest side effects.

DETAILED DESCRIPTION:
Caesarean section is associated with moderate-to-severe postoperative discomfort in a significant proportion of women, which can delay recovery and return to regular activities, disrupt mother-child bonding, affect maternal psychological well-being, and impede nursing. Furthermore, inadequate surgical pain treatment may result in hyperalgesia and chronic pain. Due to widespread misconceptions that analgesic medications or procedures may have detrimental effects on the mother or newborn, and because the severity of post-caesarean section pain is typically underestimated, pain following caesarean section is frequently under-treated.

Various analgesic therapy techniques include oral or parenteral opioids, nonsteroidal anti-inflammatory medications, and neuraxial blocks with or without adjuvants, with unclear efficacy and/or substantial adverse effects. While opioids are the gold standard for postoperative pain management, they are associated with respiratory depression, nausea, vomiting, and other adverse effects that increase patient suffering. In recent years, there has been a shift toward minimizing opioid use and developing guidelines for enhanced postpartum recovery. Studies have explored combining opioids with Nonsteroidal Anti-Inflammatory Drugs (NSAIDs), ketamine, clonidine, and dexmedetomidine for effective pain relief while avoiding opioid-related side effects.

Dexmedetomidine, a highly selective α2-agonist, is beneficial in reducing tension and anxiety. It may be effective in the management of postoperative pain due to its analgesic properties. Dexmedetomidine acts at spinal and supraspinal sites, producing antinociceptive effects via stimulation of α2-receptors in the locus coeruleus.

Ketamine has been shown to be an effective painkiller with few side effects when used in small doses. Its analgesic effects result from N-methyl-D-aspartate (NMDA) receptor antagonism, and it also interacts with opioid receptors in the brain and spinal cord. When combined with benzodiazepines, ketamine's adverse effects are further minimized.

The combination of ketamine and dexmedetomidine offers several benefits, including hemodynamic stability, absence of respiratory depression, improved postoperative analgesia, and smoother recovery. Previous work has demonstrated a synergistic effect when these agents are used together, providing excellent symptom relief while minimizing side effects.

This study seeks to address the current gap in literature regarding the comparative efficacy of different doses of dexmedetomidine combined with a fixed dose of ketamine for post-cesarean analgesia. It aims to evaluate three infusion doses of dexmedetomidine combined with ketamine using postoperative pain scores as the primary outcome measure. The findings may help optimize pain management protocols following cesarean section

ELIGIBILITY:
Inclusion Criteria:

* Elective lower segment cesarean section
* American Society of Anesthesiologists (ASA) Physical Status II
* Provided informed consent

Exclusion Criteria:

* Known drug allergy
* Presence of significant comorbidities
* Emergency surgery
* Documented psychiatric illness

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-08-16 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean Postoperative Pain Score (Visual Analog Scale) | 0-24 hours post-surgery
  Pain will be assessed using the Visual Analog Scale (VAS), a 10-point scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicate worse pain. Visual Analog Scale (VAS) scores will be recorded at 0, 2, 4, 6, 8, 12, 16, 20, and 24 hours postoperatively.

SECONDARY OUTCOMES:
Time to First Rescue Analgesia | Continuous monitoring up to 24 hours postoperative
  Measured in hours from the end of surgery to the time when the first dose of rescue analgesia (Nalbuphine 0.1 mg/kg Intravenous) is administered. Time will be recorded prospectively by anesthesia staff using standardized postoperative monitoring sheets and confirmed from the medication administration records.
Total dose of rescue analgesia (Nalbuphine) required within 24 hours | 24 hours postoperative
  Determined from direct observation and recorded in structured data collection forms by trained anesthesia personnel during the postoperative period. All doses of Nalbuphine administered will be documented in real-time and verified against the patient's medication administration records and nursing charts.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Fatima Memorial Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
VAS scores, rescue drug doses, vitals (de-identified)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication (1 year post study completion)
Access Criteria: On reasonable request by clinical researchers